CLINICAL TRIAL: NCT04431479
Title: Predicting the Quality of Response to Specific Treatments (PQRST)
Brief Title: Predicting the Quality of Response to Specific Treatments in Patients With cGVHD, PQRST Study
Status: Recruiting | Type: Observational
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: RG1006823; NCI-2020-01242 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10360 (Other: Fred Hutch/University of Washington Cancer Consortium); R01CA118953 (NIH)
Record Dates: First submitted 2020-06-11; First posted 2020-06-16 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Chronic Graft Versus Host Disease
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (questionnaire, biospecimen, chart review): Patients complete questionnaires over 10 minutes about physical symptoms, activity level, and emotional well-being and have their medical records reviewed at baseline, 1, 3, and 6 months after starting index treatment, and at start of a new systemic treatment. Patients also undergo collection of blood samples over 1-2 minutes at baseline and at 1 month after starting index treatment, or at a treatment change visit if new therapy has not started.
  Interventions: Procedure: Biospecimen Collection; Other: Medical Chart Review; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood sample
Other: Medical Chart Review — Review of medical chart
  Other Names: Chart Review
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Complete questionnaire

SUMMARY:
This trial collects clinical data and blood samples to predict the quality of response to specific treatments in patients with chronic graft-versus-host disease (cGVHD) who are about to start a new therapy. Collecting and analyzing clinical data and blood samples from patients with cGVHD before and after treatment initiation may help doctors identify changes that may predict treatment response.

DETAILED DESCRIPTION:
OUTLINE: This is an observational study.

Patients complete questionnaires over 10 minutes about physical symptoms, activity level, and emotional well-being and have their medical records reviewed at baseline, 1, 3, and 6 months after starting index treatment, and at start of a new systemic treatment. Patients also undergo collection of blood samples over 1-2 minutes at baseline and at 1 month after starting index treatment, or at a treatment change visit if new therapy has not started.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 or older
* Prior allogeneic stem cell transplant, with any graft source, donor type, and GVHD prophylaxis
* No evidence of persistent or progressive malignancy at the time of enrollment
* Agrees to be evaluated at the transplant center before a new line of treatment is started (may be concurrent with the enrollment visit), and later between 2-6 weeks, 3 months and 6 months after index treatment is started or if an additional new therapy is started before 6 months
* Signed, informed consent

Exclusion Criteria:

* Inability to comply with study procedures
* Uncontrolled psychiatric disorder
* Anticipated survival < 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic graft-versus-host disease (GVHD) who are starting a new therapy for GVHD
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-06-29 (Actual); Primary Completion 2026-08-02 (Estimated); Study Completion 2026-08-02 (Estimated)

PRIMARY OUTCOMES:
Clinical Response according to the 2014 criteria | Up to 6 months
  At the assessments, the 9 provider-reported National Institute of Health (NIH) organ severity scores (skin, eye, mouth, esophagus, upper gastrointestinal [GI], lower GI, liver, lung, and joint manifestations) will be collected reflecting disease activity in the past week. All scored items are single 4-7 point Likert scales. Based on past work, we anticipate it will take approximately 8 minutes to conduct the physical exam and record the relevant results. Pulmonary function testing results will be collected if available. Response will be assessed according to the recommendations of the 2014 NIH response measures publication or any applicable updates.
Time to next systemic treatment | From the start of the index medication until the addition of another systemic chronic graft versus host disease (cGVHD) treatment with death and treated recurrent malignancy considered competing events, assessed up to 3 years
  Any addition of another systemic cGVHD treatment for medical reasons will be considered a failure, whether added because of a new or worsening manifestation of cGVHD, used as a "steroid sparing agent," or substituted due to toxicity.
Duration of treatment | Up to 3 months
  Duration of treatment is defined as the time until discontinuation of therapeutic systemic immunosuppression (adrenal replacement and topical/local therapies are allowed) without resumption for at least 3 months.
Survival | From the start of the index medication to death with patients lost to follow up or alive at the conclusion of the study censored, assessed up to 3 years
Non-relapse mortality | Up to 3 years
  Non-relapse mortality is defined as death in remission, and relapse is considered a competing risk.
Patient-reported outcomes | Up to 3 years
  Will be assessed using Lee symptom scale and Patient Reported Outcomes Measurement Information System (PROMIS). The summary score of the Lee Symptom Scale and the PROMIS Global will be calculated according to the instructions of the developers. For analyses assessing change in quality of life, improvement or worsening of the Summary symptom score by 6 points or more or the PROMIS Physical or Mental Functioning scales by 5 points or more compared to baseline will be considered a clinically significant change.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie J. Lee, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (10):
- United States (9):
  - University of Florida, Gainesville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Dana-Farber Harvard Cancer Center, Boston, Massachusetts
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Roswell Park Cancer Institute, Buffalo, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington
- Vancouver General Hospital/BC Cancer, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hamilton BK, Onstad L, Carpenter PA, Pidala J, El Jurdi N, Farhadfar N, Kitko CL, Lee CJ, Mehta R, Chen GL, Cutler C, Lee SJ. Study Protocol: Predicting the Quality of Response to Specific Treatments (PQRST) in Chronic Graft-versus-Host Disease. Contemp Clin Trials. 2024 Oct;145:107637. doi: 10.1016/j.cct.2024.107637. Epub 2024 Jul 20. PMID 39038701